CLINICAL TRIAL: NCT03808532
Title: A Prospective Randomized Open-label Controlled Study to Assess Whether Daily Application of Skin Moisturizer Containing Acemannan Hydrogel From Birth Can Prevent Atopic Dermatitis in Children
Brief Title: Moisturizer to Prevent Atopic Dermatitis
Acronym: ACE-AD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: MYOR Ltd. (Industry)
Collaborators: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MYOR
Record Dates: First submitted 2019-01-02; First posted 2019-01-17 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Risk with Moisturizer (Experimental)
  Interventions: Other: Cura+ Moisturizing Cream
- High-Risk without Moisturizer (No Intervention)

INTERVENTIONS:
Other: Cura+ Moisturizing Cream — Parents of at-risk infants in the intervention arm will be instructed to apply moisturizer to the infant's entire body once daily for six months.
  Arms: High-Risk with Moisturizer

SUMMARY:
Atopic dermatitis (AD) is a chronic, relapsing inflammatory skin disorder associated with a decreased ability of the skin to function as an efficient immunological barrier. The disease is now two to three times more prevalent in children than it was just four decades ago. It is manifested by eczematous skin lesions associated with severe itch, leading to a significant impairment in quality of life. Of additional importance, AD oftentimes progresses to allergic rhinitis and/or asthma, a process referred to as the "atopic march." Recent reports have indicated that daily application of moisturizing creams on neonates and infants can prevent the occurrence of AD and subsequently food allergies. This is postulated to be the outcome of restoring the barrier integrity of the skin through the daily application of moisturizer.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy newborn delivered in a hospital setting more than 24 hours prior to enrollment & less than 120 hours prior to enrollment
2. Average forearm TEWL reading of >8.50 g/m2
3. Mothers must be aged >18 years
4. Parents' ability to complete questionnaire(s) at defined times throughout study duration
5. Parents or legal guardian provide informed written consent

Exclusion Criteria:

1. Preterm birth (birth prior to 37 weeks gestation)
2. Neonate has undergone major surgery or intends to undergo major surgery in the coming 14 days
3. Neonate has an existing widespread skin condition that would make the detection and/or assessment of eczema difficult
4. Neonate has been administered oral or parenteral antibiotics from birth until study enrollment
5. Neonate has a serious health issue which, at parent or investigator discretion, would make it difficult for the neonate or parents to take part in the trial
6. Any conditions which precludes the daily application of moisturizing lotion
7. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the patient safety

Ages: 24 Hours to 120 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of AD at twelve months of age in the intervention group compared to the control | 12 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema and by parental report of a medical diagnosis of AD by the infant's pediatrician and/or dermatologist

SECONDARY OUTCOMES:
Cumulative incidence of AD at six months of age in the intervention group compared to the control | 6 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema and by parental report of a medical diagnosis of AD by the infant's pediatrician and/or dermatologist
Cumulative incidence of AD at 24 months of age in the intervention group compared to the control | 24 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema and by parental report of a medical diagnosis of AD by the infant's pediatrician and/or dermatologist
Timing of onset of AD in the intervention group compared to the control | 12 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema and by parental report of a medical diagnosis of AD by the infant's pediatrician and/or dermatologist
Severity of AD in the intervention group compared to the control | 12 months
  Assessed using the Patient-Oriented Eczema Measure (POEM) questionnaire and accompanying scoring criteria. Additionally, it will be assessed by parental report of first steroidal indication by physician.
Cumulative incidence of food allergies at 12 months of age in the intervention group compared to the control | 12 months
  Evaluated with the 2010 U.S. Food and Drug Administration Food Safety Survey Questionnaire.
Cumulative incidence of food allergies at 24 months of age in the intervention group compared to the control | 24 months
  Evaluated with the 2010 U.S. Food and Drug Administration Food Safety Survey Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fridman, MD, Principal Investigator — Assuta Ashdod Hospital

IPD SHARING:
Plan to Share IPD: No